CLINICAL TRIAL: NCT04862273
Title: Native T1 Cardiac Magnetic Resonance Imaging for Diagnosis of Cardiac Amyloidosis
Brief Title: Native T1 CMR Imaging for Diagnosis of Cardiac Amyloidosis
Acronym: CMR for CA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Daniel Lavall, Cardiologist, University of Leipzig
Other Study IDs: DL-L-20006_V16
Record Dates: First submitted 2021-04-20; First posted 2021-04-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class IV; Heart Failure With Preserved Ejection Fraction; Heart Failure With Mid Range Ejection Fraction; Hypertrophy, Left Ventricular; Cardiac Amyloidosis
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Native T1 CMR: Diagnostic accuracy of native T1 CMR and ATTR probability estimator are tested against the reference methods (99mTc-DPD scintigraphy, laboratory screening for multiple myeloma / AL amyloidosis; or cardiac biopsy, if noninvasive evaluation is inconclusive)
  Interventions: Diagnostic Test: Native T1 CMR; Diagnostic Test: Web-based ATTR probability estimator (Pfizer, New York); Diagnostic Test: 99mTc-DPD scintigraphy; Diagnostic Test: Laboratory screening for multiple myeloma / AL amyloidosis; Procedure: Cardiac biopsy

INTERVENTIONS:
Diagnostic Test: Native T1 CMR — Observed method
Diagnostic Test: Web-based ATTR probability estimator (Pfizer, New York) — Observed method
Diagnostic Test: 99mTc-DPD scintigraphy — Reference method
Diagnostic Test: Laboratory screening for multiple myeloma / AL amyloidosis — Reference method
Procedure: Cardiac biopsy — If non-invasive tests for CA (99mTc-DPD scintigraphy, biochemistry) are inconclusive

SUMMARY:
The study aims to test the diagnostic accuracy of native T1 mapping for the diagnosis of cardiac amyloidosis prospectively. The hypothesis is that native T1 mapping with a cut-off value of 1341ms (3 tesla CMR) in older patients with symptomatic heart failure, increased LV wall thickness and elevated cardiac biomarkers is non-inferior to the reference method to diagnose cardiac amyloidosis (CA).

As secondary measure, a web-based ATTR probability estimator for the diagnosis of CA will be evaluated.

DETAILED DESCRIPTION:
Cardiac amyloidosis (CA) is an important differential diagnosis in older patients with symptomatic heart failure with preserved or mid-range ejection fraction and increased left ventricular wall thickness. The prevalence of CA among patients with heart failure and left ventricular (LV) hypertrophy is approximately 13%. However, diagnosis of CA is challenging because specific clinical signs are often lacking.

Amyloid fibrils deposit in the extracellular space of the myocardium increases myocardial T1 values on cardiac magnetic resonance (CMR). Therefore, native T1 imaging provides a promising non-invasive method to identify CA.

A preliminary retrospective analysis of 128 patients with increased LV wall thickness identified an area under the curve of 0.9954 (p<0.0001) for native T1 to detect CA. The optimal cut-off value was 1341ms, with a sensitivity of 100% and a specificity of 97%.

The investigators aim to test the diagnostic accuracy of native T1 mapping with the threshold of 1341ms for the diagnosis of CA compared to the reference method prospectively. Moreover, the web-based ATTR probability estimator for the diagnosis of CA will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Symptomatic heart failure (NYHA II-IV) with LVEF ≥40%
* Increased LV wall thickness (≥12mm end-diastolic)
* NT-proBNP ≥1000pg/mL
* Elevated hs-troponin T ≥14ng/L

Exclusion Criteria:

* Contraindications for CMR
* Acute myocarditis
* Acute myocardial infarction <1 month
* Severe aortic stenosis and RAISE score < 2 points

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic heart failure (NYHA functional class II to IV, LVEF ≥40%), increased left ventricular wall thickness and elevated cardiac biomarkers
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of native T1 LV mapping for diagnosis of CA | up to 7 days
  Comparison native T1 CMR with the reference method for diagnosis of CA

SECONDARY OUTCOMES:
Diagnostic accuracy of ATTR probability estimator to predict CA | up to 7 days
  Comparison of a probability score to predict ATTR with the final diagnosis of ATTR
Association of native T1 values with cardiovascular outcome | 1 years
  All-cause death, cardiovascular death and heart failure hospitalizations
Association of ATTR probability estimator values with cardiovascular outcome | 1 year
  All-cause death, cardiovascular death and heart failure hospitalizations

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided